CLINICAL TRIAL: NCT07154615
Title: Assessing Immune Dysfunction in Sepsis
Status: Not yet recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: URO-2025-34202
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ICU Patients with Sepsis
  Interventions: Other: Observational Only
- ICU Patients without Sepsis
  Interventions: Other: Observational Only
- Healthy Volunteers
  Interventions: Other: Observational Only

INTERVENTIONS:
Other: Observational Only — No intervention is included in this study

SUMMARY:
Sepsis leads to sustained immune system dysfunction resulting in increased susceptibility to secondary infection while in the hospital or after discharge. Consequently, many of the ~2 million Americans that develop sepsis every year will end up back in the ICU, weeks and months later. The objective of this study is to define the cellular and molecular mechanisms driving the dysfunction and reprogramming of T cells and B cells that mediate cellular and humoral immunity using a combination of phenotypic, functional, genomic, and metabolomic assays.

ELIGIBILITY:
ICU With Sepsis Inclusion Criteria:

* Age ≥ 18
* Presumed diagnosis of sepsis, defined as "patients with life-threatening organ dysfunction caused by a dysregulated host response to infection"
* Patients in the ICU who meet 2 or more of the quick SOFA (qSOFA) definition along with organ dysfunction:

  1. Respiration rate ≥ 22 breaths/min and/or mechanically ventilated
  2. An alteration in mental status
  3. Systolic blood pressure of less than 100 mm Hg and/or receiving inotropes to maintain blood pressure AND/OR

  <!-- -->

  1. An acute change in SOFA score ≥2 points, consequent to the infection (can assume SOFA score = 0 in patients with no pre-existing organ dysfunction)

ICU Without Sepsis Inclusion Criteria:

* Age ≥ 18
* Patients requiring care at a M Health Fairview ICU due to high acuity of illness and no other evidence of sepsis

Healthy Volunteer Inclusion Criteria

* Age greater or equal to 18
* ASA status 1, 2 or 3
* May include patients who are receiving dialysis in an outpatient setting

Exclusion Criteria (all groups):

* Active cancer with chemotherapy and/or radiation treatment within the past 6 weeks
* Medication usage that includes immunosuppressive drugs, biologic agents, cytokines, growth factor and interleukins
* Steroid medication usage of > 300mg hydrocortisone per day (equivalent of > 20mg prednisone). Patients with chronic steroid use will be excluded, however patients who have had stress dose steroids administered following admission will be included.
* Patients with a history of, or who currently have evidence of autoimmune disease, including but not limited to: myasthenia gravis, Guillain Barré syndrome, systemic lupus erythematosus, multiple sclerosis, scleroderma, ulcerative colitis, Crohn's disease, autoimmune hepatitis, Wegener's granulomatosis, HIV/AIDS, etc.
* Patients with active or a history of acute or chronic lymphocytic leukemia
* Known history of chronic hepatitis B (HBV) infection and not on treatment with HBV nucleoside analogues prior to the current hospitalization, or HBV DNA > 100 IU/mL
* Known history of infection with hepatitis C (HCV) and currently undergoing treatment for HCV infection or has detectable HCV RNA
* Participation in another investigational interventional drug study within the past 4 weeks
* Current pregnancy
* Current incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with and without sepsis in the ICU, compared to healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
EliSpot - Day 1 | Day 1
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
EliSpot - Day 4 | Day 4
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
EliSpot - Day 7 | Day 7
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
EliSpot - Day 14 | Day 14
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
EliSpot - Day 21 | Day 21
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
EliSpot - Day 28 | Day 28
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Ex Vivo TNF Production - Day 1 | Day 1
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Ex Vivo TNF Production - Day 4 | Day 4
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Ex Vivo TNF Production - Day 7 | Day 7
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Ex Vivo TNF Production - Day 14 | Day 14
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Ex Vivo TNF Production - Day 21 | Day 21
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Ex Vivo TNF Production - Day 28 | Day 28
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Flow Cytometry of Peripheral Blood Leukocytes - Day 1 | Day 1
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Flow Cytometry of Peripheral Blood Leukocytes - Day 4 | Day 4
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Flow Cytometry of Peripheral Blood Leukocytes - Day 7 | Day 7
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Flow Cytometry of Peripheral Blood Leukocytes - Day 14 | Day 14
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Flow Cytometry of Peripheral Blood Leukocytes - Day 21 | Day 21
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Flow Cytometry of Peripheral Blood Leukocytes - Day 28 | Day 28
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Quantification of Cytokines in Serum - Day 1 | Day 1
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Quantification of Cytokines in Serum - Day 4 | Day 4
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Quantification of Cytokines in Serum - Day 7 | Day 7
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Quantification of Cytokines in Serum - Day 14 | Day 14
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Quantification of Cytokines in Serum - Day 21 | Day 21
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Quantification of Cytokines in Serum - Day 28 | Day 28
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Quantification of Chemokines in Serum - Day 1 | Day 1
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Quantification of Chemokines in Serum - Day 4 | Day 4
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Quantification of Chemokines in Serum - Day 7 | Day 7
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Quantification of Chemokines in Serum - Day 14 | Day 14
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Quantification of Chemokines in Serum - Day 21 | Day 21
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Quantification of Chemokines in Serum - Day 28 | Day 28
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Transcriptional Profiling - Day 1 | Day 1
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Transcriptional Profiling - Day 4 | Day 4
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Transcriptional Profiling - Day 7 | Day 7
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Transcriptional Profiling - Day 14 | Day 14
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Transcriptional Profiling - Day 21 | Day 21
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
Transcriptional Profiling - Day 28 | Day 28
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
CBC - Day 1 | Day 1
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
CBC - Day 4 | Day 4
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
CBC - Day 7 | Day 7
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
CBC - Day 14 | Day 14
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
CBC - Day 21 | Day 21
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes
CBC - Day 28 | Day 28
  Sample analysis to determine waxing and waning of Course of Sepsis parameters associated with clinical outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Griffith, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No